CLINICAL TRIAL: NCT03936842
Title: Evaluation of an Educational Intervention for Women With Breast Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CCR5063
Record Dates: First submitted 2019-04-18; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Breast Pain; Mastalgia
MeSH Terms: conditions — Mastodynia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Eligible patients who are referred to the "one-stop" diagnostic clinic with breast pain alone and have completed a clinical assessment will be given a patient information sheet inviting them to participate in the study. They will be met by the interviewing clinician at the same visit.
  Interventions: Behavioral: Breast Pain video; Behavioral: Semi-structure interviews

INTERVENTIONS:
Behavioral: Breast Pain video — An educational video of approximately 10 minutes about breast pain, self-examination and breast awareness will be shown to the participant.
Behavioral: Semi-structure interviews — A semi-structured, face-to-face interview will be then undertaken. The principles of Grounded Theory will be used to guide the interview. All of the interviews will be recorded and transcribed securely, only referencing the patient according to their study number. Their name and hospital number will not be used.

SUMMARY:
Evaluation of an educational intervention for women with breast pain

Target Problem -Symptomatic breast pain Study Objectives- The primary objective is to obtain knowledge of women's perceptions of an educational video about breast pain, breast awareness and self-examination and its impact on their confidence in self-management of breast pain.

The secondary objectives -proportion of women who report that the video

1. Was informative
2. Might have reassured them enough not to have needed to seek an appointment in secondary care.

Study Design- Prospective single-centre mixed methods study through semi-structured interviews for Masters in Public Health thesis Trial Population -Women, aged 18-40, referred to "one-stop" / rapid diagnostic breast clinic at The Royal Marsden Hospital (RMH) with breast pain alone.

Recruitment target Until saturation, expected sample 10-15 Trial Design- Mixed methods study using semi-structured interviews Primary endpoint -This is a qualitative study, with no statistical primary end point.

Secondary endpoints-Descriptive summaries of two questions will be reported as a secondary end point.

Inclusion Criteria

* Women aged between 18 years and 40 years on the day of clinic attendance
* Breast pain as the only symptom
* Normal clinical examination
* No further investigation (imaging, biopsy etc) Exclusion Criteria
* Presence of suspicious features during clinical examination requiring further investigation
* Strong family history of breast cancer
* Previous breast imaging within last 12 months
* Previous history of breast cancer
* Current or previous treatment with Tamoxifen
* Concurrent cancer
* Medical or psychiatric illness which might impact their participation in the study

DETAILED DESCRIPTION:
The prevalence of breast pain has been reported to be between 41-69% in clinical cohorts and in the general population (1-4). The incidence of cancer in women with breast pain alone (ie no lump or other, more concerning symptoms) is low, with published rates between 1 to 1.8% (7-9).

Furthermore, the prevalence of breast pain increases linearly up to the age of 50 and then decreases (4), thus women under 40 with a normal clinical examination do not require further investigations and can be reassured in primary care.

Despite this, mastalgia is one of the most common symptoms in women referred to a breast unit representing up to 69% of attendances (5-7). Consequently, women affected by breast pain are up to 4.7 times more likely to have had a mammogram than asymptomatic women (6). ln order to facilitate early breast cancer diagnosis there is a suspected cancer pathway referral (for an appointment within 2 weeks) from primary care to specialist units. Recent increases in breast urgent referrals have increased the pressure on already overstretched services.

Many strategies have been tried to manage the tension between the desire for early detection of breast cancer, and avoiding unnecessary referral for normal breast sensations.

Although breast screening by self-examination or clinical examination has not been shown to reduce breast cancer mortality in studies (10), breast awareness can be linked to early detection that facilitates treatment and has the potential to reduce mortality (11). Therefore, breast awareness and self-examination have become relevant parts of general breast education promoting women's confidence to discern between normality and unusual changes (12-17). Self-examination is not frequently taught in primary care and "there is a need to develop more innovative strategies to promote breast health awareness and early detection of breast cancer in women" (18). In this study, as part of a Masters in Health Policy, we are investigating the impact of an educational video, here to be shown after a clinic appointment, but with the potential to be distributed to general practitioners, and to patients directly if favourably received.

Methodology

1. Patient recruitment 1.1 Initial visit to "one-stop"clinic Eligible patients who are referred to the "one-stop" diagnostic clinic with breast pain alone and have completed a clinical assessment will be given a patient information sheet inviting them to participate in the study. They will be met by the interviewing clinician at the same visit.

   1.2 Consent Consent will be sought by the clinician who will undertake the interviews.
2. Intervention: educational video An educational video of approximately 10 minutes about breast pain, self-examination and breast awareness will be shown to the participant.
3. Semi-structured interview A semi-structured, face-to-face interview will be then undertaken. The principles of Grounded Theory will be used to guide the interview. All of the interviews will be recorded and transcribed securely, only referencing the patient according to their study number. Their name and hospital number will not be used.

A number of pre-planned, open questions will be asked. The core questions are related to the topic of discussion - impressions related to the intervention and subsequent effect into their previous concerns. Further questions will evolve in response to answers given by earlier participants. The duration of the interview will depend on the extent of the answers and any follow-up questions that derive later from earlier answers.

Data Acquisition and analysis The video show and interview will be undertaken in a private room after routine clinical assessment. The interviewer will be the MSc student, a medically-qualified breast clinician with an interest in breast pain, who has read the relevant literature. The recorded interview and notes taken by investigator during the interview are the only data.

The analysis will run alongside data collection as an iterative process to inform further sampling. The purpose of the analysis is to describe the participants' opinion and to develop theoretical explanations for these. The interviews will be analysed by reading the transcripts in detail and assigning codes to give meaning to segments of the text. Emerging codes will be grouped into themes and discussed and then explored in subsequent interviews. The analysis will be undertaken using the constant comparison technique of grounded theory whereby data will be examined for differences and similarities within the themes, taking into account the patient context. The initial codes will be modified and new codes added as the project progresses. New data will be compared with previous interviews to identify the similarities and differences.

Evaluation of Outcome This is a mixed methods study. As a result, we will have increased knowledge of the perceptions of women presenting with breast pain about an educational video. We will have some quantitative information about whether they find it informative and whether it might lead them to avoid attending secondary care. It will guide the future management of women with pain at the interface of primary and secondary care.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female patients aged between 18 years and 40 years on the day of clinic attendance (referred to one-stop breast clinic with breast pain alone)
* Normal examination in clinic
* No further breast investigations undertaken or required

Exclusion Criteria:

* Presence of concerning features during clinical examination requiring further investigation
* Pregnancy or lactation at the time of study diagnosis.
* Strong family history of breast cancer
* Recent previous imaging or clinic attendance for same symptom within last 12 months
* Previous history of breast cancer
* Current or previous treatment with Tamoxifen
* Medical or psychiatric illness which, in the opinion of the assessing clinician, might impact their participation in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Estimated)
Dates: Start 2019-05-31 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient's perceptions on the breast-pain video | 10 minutes
  Due to the semi-structure interview qualitative nature of the study the primary objective is to obtain observational data for insights and patterns (through "quotes") of women's perceptions of an educational video about breast pain, breast awareness and self-examination and its impact on their confidence in self-management of breast pain.

SECONDARY OUTCOMES:
Video's purpose evaluation | 10 minutes
  proportion of women who report that the video
  1. Was informative
  2. Might have reassured them enough not to have needed to seek an appointment in secondary care

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ader DN, Shriver CD. Update on clinical and research issues in cyclical mastalgia. Breast J 1998;4:25-32.
- [Background] Boyle CA, Berkowitz GS, Kelsey JL. Epidemiology of premenstrual symptoms. Am J Public Health. 1987 Mar;77(3):349-50. doi: 10.2105/ajph.77.3.349. PMID 3812845
- [Background] Smith RL, Pruthi S, Fitzpatrick LA. Evaluation and management of breast pain. Mayo Clin Proc. 2004 Mar;79(3):353-72. doi: 10.4065/79.3.353. PMID 15008609
- [Background] Scurr J, Hedger W, Morris P, Brown N. The prevalence, severity, and impact of breast pain in the general population. Breast J. 2014 Sep-Oct;20(5):508-13. doi: 10.1111/tbj.12305. Epub 2014 Jul 7. PMID 25041468
- [Background] Newton P, Hannay DR, Laver R. The presentation and management of female breast symptoms in general practice in Sheffield. Fam Pract. 1999 Aug;16(4):360-5. doi: 10.1093/fampra/16.4.360. PMID 10493705
- [Background] Ader DN, Browne MW. Prevalence and impact of cyclic mastalgia in a United States clinic-based sample. Am J Obstet Gynecol. 1997 Jul;177(1):126-32. doi: 10.1016/s0002-9378(97)70450-2. PMID 9240595
- [Background] Barton MB, Elmore JG, Fletcher SW. Breast symptoms among women enrolled in a health maintenance organization: frequency, evaluation, and outcome. Ann Intern Med. 1999 Apr 20;130(8):651-7. doi: 10.7326/0003-4819-130-8-199904200-00005. PMID 10215561
- [Background] Eberl MM, Phillips RL Jr, Lamberts H, Okkes I, Mahoney MC. Characterizing breast symptoms in family practice. Ann Fam Med. 2008 Nov-Dec;6(6):528-33. doi: 10.1370/afm.905. PMID 19001305
- [Background] Joyce DP, Alamiri J, Lowery AJ, Downey E, Ahmed A, McLaughlin R, Hill AD. Breast clinic referrals: can mastalgia be managed in primary care? Ir J Med Sci. 2014 Dec;183(4):639-42. doi: 10.1007/s11845-013-1066-z. Epub 2014 Jan 9. PMID 24402166
- [Background] Kosters JP, Gotzsche PC. Regular self-examination or clinical examination for early detection of breast cancer. Cochrane Database Syst Rev. 2003;2003(2):CD003373. doi: 10.1002/14651858.CD003373. PMID 12804462
- [Background] Richards MA. The National Awareness and Early Diagnosis Initiative in England: assembling the evidence. Br J Cancer. 2009 Dec 3;101 Suppl 2(Suppl 2):S1-4. doi: 10.1038/sj.bjc.6605382. PMID 19956152
- [Background] Mac Bride MB, Pruthi S, Bevers T. The evolution of breast self-examination to breast awareness. Breast J. 2012 Nov-Dec;18(6):641-3. doi: 10.1111/tbj.12023. Epub 2012 Sep 26. No abstract available. PMID 23009674
- [Background] Byrne S, Robles-Rodriguez E. Educational parties as a strategy to promote breast health awareness and screening in underserved female populations. Oncol Nurs Forum. 2009 Mar;36(2):145-8. doi: 10.1188/09.ONF.145-148. No abstract available. PMID 19273403
- See also: National Institute for Health and Clinical Excellence (NICE). Familial Breast Cancer: Full Guideline. — https://www.nice.org.uk/guidance/cg164
- See also: International Agency for Research on Cancer (IARC). IARC Screening Group. — http://screening.iarc.fr/breastselfexamination.php
- See also: National Office of NHS Cancer Screening Programmes, Public Health England. NHS Breast Cancer Screening Programme 2013 — http://www.cancerscreening.nhs.uk/breastscreen/breastawareness.html